CLINICAL TRIAL: NCT04856176
Title: A Phase II Trial of GM-CSF Plus Maintenance Pembrolizumab +/- Pemetrexed After Completion of First Line Chemo-Immunotherapy in Advanced Non-Small Cell Lung Cancer Patients with PDL-1 of 1%-49%
Brief Title: A Study of Sargramostim Plus Pembrolizumab with or Without Pemetrexed in Patients with Advance Non-small Cell Lung Cancer After Completion of Chemoimmunotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Tufts Medical Center (Other)
Collaborators: Partner Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GM-CSF
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Non-Small Cell Carcinoma of Lung, TNM Stage 4
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; pembrolizumab; Pemetrexed; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: This is a Phase II open-label, single-center, single arm trial using a Simon two-stage optimal design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GM-CSF Plus Maintenance Pembrolizumab +/- Pemetrexed (Experimental): All patients will receive GM-CSF plus maintenance pembrolizumab with or without pemetrexed, following completion of 4 cycles of chemo-immunotherapy
  Interventions: Drug: Granulocyte-Macrophage Colony-Stimulating Factor; Drug: Pembrolizumab; Drug: pemetrexed; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Granulocyte-Macrophage Colony-Stimulating Factor — 250 mcg
Drug: Pembrolizumab — 200mg every 3 weeks
Drug: pemetrexed — 500mg/m2
Drug: Paclitaxel — 200mg/m2
Drug: Carboplatin — AUC 5/6

SUMMARY:
Metastatic lung cancer is the leading cause of cancer mortality worldwide with a 5-year survival of less than 5%. With the approval of programmed cell death 1 (PD-1) inhibitors in advanced lung cancer, such as pembrolizumab, there has been an improvement in overall response rates (ORR) and survival compared to chemotherapy.

However, there is still a need for improvement in response rates in first-line treatments for patients with stage 4 NSCLC without genetically targetable alterations, especially in those patients with PDL-1 <50%.

This trial is important because it seeks to discover whether the responses seen in first line treatments with PD-1 inhibitors + chemotherapy can be augmented with the addition of GM-CSF during the maintenance phase with pembrolizumab +/- pemetrexed.

DETAILED DESCRIPTION:
Lung cancer is the most commonly diagnosed cancer worldwide. Metastatic lung cancer is the leading cause of cancer mortality worldwide with a 5-year survival of less than 5%. With the approval of programmed cell death 1 (PD-1) inhibitors in advanced lung cancer, there has been an improvement in overall response rates and survival compared to chemotherapy.

Checkpoint inhibition has become a primary treatment modality for vast number of cancers including lung cancer, prolonging survival in some patients. However, an important consideration is how to best select those patients who will respond to checkpoint inhibition. The biomarker that has been studied most extensively is PD-L1 expression. Studies have shown trends for increased response rates to PD-1 blockade in PD-L1 positive tumors.

NSCLC patients are now approved for pembrolizumab monotherapy (PDL-1>1%) or for pembrolizumab in combination with chemotherapy (carboplatin/pemetrexed for non-squamous or carboplatin/paclitaxel) (no minimum PDL-1). As the ORR and PFS in both these trials indicate, however, there is a need for improvement in response rates and PFS in first-line treatments for patients with stage 4 NSCLC without genetically targetable alterations especially in those patients with PDL-1 <50%.

There are both pre-clinical and clinical evidence supporting the combination of granulocyte macrophage colony stimulating factor (GM-CSF) with immunotherapy. GM-CSF is a hematopoietic growth factor that triggers proliferation and differentiation of hematopoietic progenitor cells, mainly neutrophils, monocytes/macrophages and myeloid-derived dendritic cells, and is approved by the FDA for this purpose.

A phase II randomized clinical trial of unresectable stage III or IV melanoma patients comparing the effects of ipilimumab plus GM-CSF vs ipilimumab alone was shown to be both safe and had longer overall survival with lower toxicity than immunotherapy alone; 1 year survival for ipilimumab plus sargramostim was 68.9% (95% CI, 60.6%-85.5%) compared to 52.9% (95% CI, 43.6%-62.2%) for ipilimumab alone.

It is hypothesized that the use of GM-CSF along with a PD-1 inhibitor +/- pemetrexed is safe and will increase the overall response rate and progression-free survival in advanced NSCLC patients with PDL-1 of 1%-49%. This will establish the basis for further evaluation of GM-CSF+PD-1 in advanced NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Histologically confirmed stage 4 NSCLC or stage 3B/3C not able to receive chemoradiation with no sensitizing EGFR or ALK mutations.
3. PDL-1 of 1%-49%
4. No previous history of immunotherapy treatment
5. ECOG PS 0-1
6. At least one measurable lesion according to RECIST version 1.1
7. Life expectancy of at least 3 months.
8. Able to self-administer daily GM-CSF injections
9. Eligible for treatment with 4 cycles of chemoimmunotherapy followed by maintenance therapy with pembrolizumab +/- pemetrexed.

Exclusion Criteria:

1. Receiving systemic glucocorticoids or other immunosuppressive treatment
2. Untreated brain metastases
3. Active autoimmune disease
4. Active interstitial lung disease, pneumonitis
5. Solid organ transplant recipients
6. Subject may not participate in another drug research study while participating in this research study
7. Pregnant patients
8. Known hypersensitivity to GM-CSF (sargramostim)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 24 Months
  Progression is measured according to RECIST 1.1 criteria.
Overall Survival (OS) | 24 months
  Patient survival status throughout their participation in the study

SECONDARY OUTCOMES:
To evaluate changes in monocytes at different time points during study treatment | 24 Months
  Time points include study weeks 0, 12, 14 and 15
To evaluate changes in myeloid derived suppressor cells at different time points during study treatment | 24 Months
  Time points include study weeks 0, 12, 14 and 15
To evaluate changes in CD4 T at different time points during study treatment | 24 Months
  Time points include study weeks 0, 12, 14 and 15
To evaluate changes in CD8 T at different time points during study treatment | 24 Months
  Time points include study weeks 0, 12, 14 and 15
To evaluate changes in PD-1+ CD4 at different time points during study treatment | 24 Months
  Time points include study weeks 0, 12, 14 and 15
To evaluate changes in PD-1+ CD8 at different time points during study treatment | 24 Months
  Time points include study weeks 0, 12, 14 and 15

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- [Background] Paz-Ares L, Luft A, Vicente D, Tafreshi A, Gumus M, Mazieres J, Hermes B, Cay Senler F, Csoszi T, Fulop A, Rodriguez-Cid J, Wilson J, Sugawara S, Kato T, Lee KH, Cheng Y, Novello S, Halmos B, Li X, Lubiniecki GM, Piperdi B, Kowalski DM; KEYNOTE-407 Investigators. Pembrolizumab plus Chemotherapy for Squamous Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Nov 22;379(21):2040-2051. doi: 10.1056/NEJMoa1810865. Epub 2018 Sep 25. PMID 30280635
- [Background] Shi X, Zhang X, Li J, Mo L, Zhao H, Zhu Y, Hu Z, Gao J, Tan W. PD-1 blockade enhances the antitumor efficacy of GM-CSF surface-modified bladder cancer stem cells vaccine. Int J Cancer. 2018 May 15;142(10):2106-2117. doi: 10.1002/ijc.31219. Epub 2017 Dec 26. PMID 29243219
- [Background] Hodi FS, Butler M, Oble DA, Seiden MV, Haluska FG, Kruse A, Macrae S, Nelson M, Canning C, Lowy I, Korman A, Lautz D, Russell S, Jaklitsch MT, Ramaiya N, Chen TC, Neuberg D, Allison JP, Mihm MC, Dranoff G. Immunologic and clinical effects of antibody blockade of cytotoxic T lymphocyte-associated antigen 4 in previously vaccinated cancer patients. Proc Natl Acad Sci U S A. 2008 Feb 26;105(8):3005-10. doi: 10.1073/pnas.0712237105. Epub 2008 Feb 19. PMID 18287062
- [Background] Fong L, Kwek SS, O'Brien S, Kavanagh B, McNeel DG, Weinberg V, Lin AM, Rosenberg J, Ryan CJ, Rini BI, Small EJ. Potentiating endogenous antitumor immunity to prostate cancer through combination immunotherapy with CTLA4 blockade and GM-CSF. Cancer Res. 2009 Jan 15;69(2):609-15. doi: 10.1158/0008-5472.CAN-08-3529. PMID 19147575
- [Background] Nemunaitis, J., Schiller, H., Ross, H., et. al. A Phase 2 Randomized Study of GM-CSF Gene-Modified Autologous Tumor Cell Immunotherapy (CG8123) with and without Low-Dose Cyclophosphamide in Advanced Stage Non-Small Cell Lung Cancer (NSCLC). Molecular Therapy 2006; Volume 13, Supplement 1
- [Background] Hodi FS, Lee S, McDermott DF, Rao UN, Butterfield LH, Tarhini AA, Leming P, Puzanov I, Shin D, Kirkwood JM. Ipilimumab plus sargramostim vs ipilimumab alone for treatment of metastatic melanoma: a randomized clinical trial. JAMA. 2014 Nov 5;312(17):1744-53. doi: 10.1001/jama.2014.13943. PMID 25369488
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835
- [Background] Kwek SS, Kahn J, Greaney SK, Lewis J, Cha E, Zhang L, Weber RW, Leonard L, Markovic SN, Fong L, Spitler LE. GM-CSF and ipilimumab therapy in metastatic melanoma: Clinical outcomes and immunologic responses. Oncoimmunology. 2015 Oct 29;5(4):e1101204. doi: 10.1080/2162402X.2015.1101204. eCollection 2016 Apr. PMID 27141383
- [Background] Ohradanova-Repic A, Machacek C, Fischer MB, Stockinger H. Differentiation of human monocytes and derived subsets of macrophages and dendritic cells by the HLDA10 monoclonal antibody panel. Clin Transl Immunology. 2016 Jan 8;5(1):e55. doi: 10.1038/cti.2015.39. eCollection 2016 Jan. PMID 26900469
- [Background] Soiffer R, Lynch T, Mihm M, Jung K, Rhuda C, Schmollinger JC, Hodi FS, Liebster L, Lam P, Mentzer S, Singer S, Tanabe KK, Cosimi AB, Duda R, Sober A, Bhan A, Daley J, Neuberg D, Parry G, Rokovich J, Richards L, Drayer J, Berns A, Clift S, Cohen LK, Mulligan RC, Dranoff G. Vaccination with irradiated autologous melanoma cells engineered to secrete human granulocyte-macrophage colony-stimulating factor generates potent antitumor immunity in patients with metastatic melanoma. Proc Natl Acad Sci U S A. 1998 Oct 27;95(22):13141-6. doi: 10.1073/pnas.95.22.13141. PMID 9789055
- [Background] Scagliotti GV, Parikh P, von Pawel J, Biesma B, Vansteenkiste J, Manegold C, Serwatowski P, Gatzemeier U, Digumarti R, Zukin M, Lee JS, Mellemgaard A, Park K, Patil S, Rolski J, Goksel T, de Marinis F, Simms L, Sugarman KP, Gandara D. Phase III study comparing cisplatin plus gemcitabine with cisplatin plus pemetrexed in chemotherapy-naive patients with advanced-stage non-small-cell lung cancer. J Clin Oncol. 2008 Jul 20;26(21):3543-51. doi: 10.1200/JCO.2007.15.0375. Epub 2008 May 27. PMID 18506025
- [Background] Kaplan D, Sun Z, Tallman MS, Flinn IW, Xiao W, Caimi PF, Kaye NM, Lazarus HM. Prognostic information and biological insights in chronic lymphocytic leukemia by high-resolution immunophenotypic analysis of ZAP70. Cytometry A. 2014 Sep;85(9):798-808. doi: 10.1002/cyto.a.22485. Epub 2014 May 20. PMID 24845539
- [Background] Kaplan D, Smith D. Enzymatic amplification staining for flow cytometric analysis of cell surface molecules. Cytometry. 2000 May 1;40(1):81-5. doi: 10.1002/(sici)1097-0320(20000501)40:13.0.co;2-k. PMID 10754521
- [Background] Kaplan D, Smith D, Meyerson H, Pecora N, Lewandowska K. CD5 expression by B lymphocytes and its regulation upon Epstein-Barr virus transformation. Proc Natl Acad Sci U S A. 2001 Nov 20;98(24):13850-3. doi: 10.1073/pnas.241509398. Epub 2001 Nov 13. PMID 11707593
- [Background] Lazarus HM, Sommers SR, Arfons LM, Fu P, Ataergin SA, Kaye NM, Liu F, Kindwall-Keller TL, Cooper BW, Laughlin MJ, Creger RJ, Barr PM, Gerson SL, Kaplan D. Spontaneous autologous graft-versus-host disease in plasma cell myeloma autograft recipients: flow cytometric analysis of hematopoietic progenitor cell grafts. Biol Blood Marrow Transplant. 2011 Jul;17(7):970-8. doi: 10.1016/j.bbmt.2011.03.005. Epub 2011 Apr 11. PMID 21440080